CLINICAL TRIAL: NCT07076290
Title: A Repeat Ascending Dosing Study of the Safety and Clinical Activity of R-3750 in Patients With Mild to Moderate COPD
Acronym: R-3750-01-LU
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rise Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RISE-3750-01LU
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); COPD Exacerbation; COPD Exacerbation Acute
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label R-3750 (Other): Open Label Drug - R-3750
  Interventions: Drug: R-3750

INTERVENTIONS:
Drug: R-3750 — R-3750 DP; Lactococcus lactis expressing Surface Layer Protein A (SlpA)

SUMMARY:
The goal of this study is to determine the safety and tolerability of orally taken probiotic (R-3750) in patients with mild to moderate chronic obstructive pulmonary disease (COPD)

DETAILED DESCRIPTION:
Patients will take an oral dosage of probiotic (R-3750) and provide patient-reported and scored measure of their chronic obstructive pulmonary disease (COPD). Blood and fecal evaluations of inflammation and assessment of probiotic (R-3750) on fecal levels will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinically documented history of COPD for at least 1 year in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Subjects must present with the following: a measured pre and post-salbutamol Forced expiratory volume in one second/ Forced vital capacity (FEV1/FVC) ratio of <0.70 to confirm the diagnosis of COPD; a measured post-salbutamol FEV1>20% and ≤80% of predicted normal values
* Baseline mMRC dyspnea score 1 to 3
* Post-bronchodilator FEV1 > 50% predicted (GOLD COPD grade 1-2)
* Smoking pack years ≥ 10 years
* Age ≥ 40 years
* Acceptable standard-of-care COPD maintenance therapy includes long-acting beta-agonists (LABAs), long-acting muscarinic antagonists (LAMAs), inhaled corticosteroids (ICS), or combinations thereof (e.g., dual LABA/LAMA, or triple LABA/LAMA/ICS therapy). The patient must have been on a stable dose and regimen for at least 4 weeks prior to screening with no changes anticipated during the study unless medically necessary.
* A history of ≥ 1 exacerbations in the last 12 months
* Be able to provide written consent; compliant with study procedures and study visits.

Exclusion Criteria:

* Patients whose treatment is considered palliative (life expectancy <12 months) Comorbid severe lung disease, such as bronchiectasis, pulmonary fibrosis
* Current smoker or cessation within 3 months of screening, or current use of vaping device
* Patients with pneumonia or COPD exacerbation or lower respiratory infections within the 4 weeks prior to study Day 1
* Uncontrolled co-morbid conditions, such as diabetes mellitus, hypertension and heart failure [e.g. New York Heart Association (NYHA) class III (e.g. less than ordinary activity causes fatigue, palpitation, or dyspnea), and class IV (e.g. Symptoms of heart failure at rest)] that will affect the study.
* Myocardial infarction, unstable angina or stroke within 12 months prior to screening
* Diagnosis of malignancy within 5 years of study Day 1(except for excised localized carcinoma of skin not including malignant melanoma)
* Clinically significant ECG changes, which in the opinion of investigator warrants further investigations
* Evidence of alcohol, drug or solvent abuse.
* Pregnant, breastfeeding, or lactating women. Women of child-bearing potential (i.e. not surgically sterilized or post- menopausal) must have a negative blood serum pregnancy test performed at the screening visit and must agree to use two methods of birth control (one of which must be a barrier method) for at least 3 months past the last day on the study.
* Participation in an interventional clinical study within 3 months of study Day 1 or receipt of any investigational medicinal product within 3 months or 5 half- lives.
* Lung volume reduction surgery or bronchoscopic lung volume reduction within the last 12 months.
* Historical or current evidence of clinically significant neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Other conditions that could lead to elevated eosinophils such as Hypereosinophilic syndromes including Eosinophilic Granulomatosis with Polyangiitis, or Eosinophilic Esophagitis.
* Cirrhosis or current unstable liver disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice. Stable noncirrhotic chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B or C -e.g., presence of hepatitis B surface antigen [HbsAg] or positive hepatitis C antibody test result) is acceptable if the participant otherwise meets entry criteria.
* Active blood born infection (e.g. HIV, Hepatitis A, B or C)
* Current or recent (<2 weeks) treatment with oral steroids, theophylline, chronic azithromycin or other methylxanthines, roflumilast, or Dupixent
* Current infection or antibiotic treatment
* Use of probiotics within 2 weeks of study Day 1
* Subjects with a current diagnosis of asthma (those with a prior history are eligible if they meet inclusion criteria for a current diagnosis of COPD)
* Subjects receiving treatment with oxygen more than 4.0 Litres/minute (L/min). While breathing supplemental oxygen, subjects should demonstrate oxyhemoglobin saturation greater than or equal to 89 percent.

Ages: 40 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the treatment-related adverse events of R-3750 | 12 weeks
  To assess the number of participants with treatment-related adverse events after taking R-3750 (probiotics)

SECONDARY OUTCOMES:
Clinical Response based on St. George's Respiratory Questionnaire (SGRQ) | 12 weeks
  To assess the number of participants that show improvements in the chronic obstructive pulmonary disease (COPD) severity by collecting the St. George's Respiratory Questionnaire (SGRQ). The scores are based on a numbering system ranging from 0-100 where the higher number indicates a worse condition. The scores will be compared from the beginning of the trial and again at different times to the end to see if there are any changes in symptoms before and after taking R-3750 (probiotic).

IPD SHARING:
Plan to Share IPD: No